CLINICAL TRIAL: NCT07066904
Title: Quantification of Mitral Regurgitation Using 4D MRI Flow : Comparison With 2D MRI Flow and Echocardiography Using the Evolution of Left Ventricular Remodeling as a Reference
Acronym: FLAME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); GIRCI IDF (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP240794; PHRCI-2023-45 (Other Grant/Funding Number: French ministry of health); 2024-A01894-43 (Other: Agence nationale de sécurité du médicament et des produits de santé); 25.00001.000350 (Other: Commission Nationale des Recherche Impliquant la Personne Humaine)
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Mitral Regurgitation (MR)
Keywords: Mitral regurgitation; 4D MRI; 4D-flow MRI; cardiovascular magnetic resonance; Ultrafast ultrasound imaging; ultrafast echocardiography
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild mitral regurgitation (Experimental): Patient suffuring from mild mitral regurgitation (n=30)
  Interventions: Diagnostic Test: Standard echocardiography; Diagnostic Test: 2D phase-contrast magnetic resonance imaging; Diagnostic Test: 4D flow magnetic resonance imaging; Diagnostic Test: Cardiac ultrafast ultrasound imaging
- Moderate mitral regurgitation (Experimental): Patient suffuring from moderate mitral regurgitation (n=30)
  Interventions: Diagnostic Test: Standard echocardiography; Diagnostic Test: 2D phase-contrast magnetic resonance imaging; Diagnostic Test: 4D flow magnetic resonance imaging; Diagnostic Test: Cardiac ultrafast ultrasound imaging
- Severe mitral regurgitation (Experimental): Patient suffuring from severe mitral regurgitation (n=100)
  Interventions: Diagnostic Test: Standard echocardiography; Diagnostic Test: 2D phase-contrast magnetic resonance imaging; Diagnostic Test: 4D flow magnetic resonance imaging; Diagnostic Test: Cardiac ultrafast ultrasound imaging

INTERVENTIONS:
Diagnostic Test: Standard echocardiography — Routine ultrasound examination with standardized recordings for the study, incorporating volumetric assessment techniques
  Other Names: Cardiac echography; TTE; Heart ultrasounds
Diagnostic Test: 2D phase-contrast magnetic resonance imaging — A cardiac MRI will be performed on a 1.5 Tesla system, including a biventricular function study with a series of short-axis slices, three long-axis slices, a 2D phase-contrast acquisition orthogonal to the aortic root. Additionally, standard T1 mapping sequences will be acquired on three short-axis slices, 15 minutes after the injection of 0.2 mmol/kg of body weight of gadolinium, for myocardial and blood T1 measurements.
  Other Names: 2D MRI; Cardiac magnetic resonance imaging; CMR
Diagnostic Test: 4D flow magnetic resonance imaging — A sagittal 4D flow acquisition lasting between 6 and 10 minutes of free breathing to cover all four cardiac chambers is added to the 2D acquisition.
  Other Names: 4D MRI
Diagnostic Test: Cardiac ultrafast ultrasound imaging — Ultrafast sequences are added to the standard echocardiography acquisition.
  Other Names: ultrafast echocardiography

SUMMARY:
The goal of this study is to evaluate whether 4D MRI provides a better assessment of mitral regurgitation quantification and associated ventricular remodeling than standard imaging techniques: echocardiography and 2D MRI, in patients suffuring from mitral regurgitation. 4D MRI demonstrated its superiority to 2D MRI in some other valve diseases but remains not widely used, due to a lack of evidence. The main question our study aims to answer is:

• Is mitral regurgitant volume measured on 4D MRI more strongly related to remodeling progression (after correction of regurgitation or not) than regurgitant volume measured on 2D MRI and echocardiography?

Participants will undergo 4D MRI, 2D MRI and echocardiography twice at six-month intervals.

DETAILED DESCRIPTION:
Mitral Regurgitation (MR) is a widely prevalent valvular disease. The decision to refer patients for intervention relies on the precise quantification of MR using the mitral regurgitant volume. This quantification is primarily performed through transthoracic echocardiography (TTE), but its accuracy is limited by operator dependency and acoustic windows.

Magnetic resonance imaging (MRI) is now considered the preferred alternative technique for measuring mitral regurgitant volume using 2D phase-contrast sequences. However, it requires significant expertise from specialized centers.

4D flow MRI enables the recording of blood flow velocities in all directions across the entire cardiac volume and has demonstrated superiority over 2D MRI in other valvular diseases. However, limited data are available for validating the estimation of mitral regurgitation using 4DFlow-MRI, mainly due to the absence of a reference technique. As previously proposed for comparisons between 2D MRI and TTE, ventricular remodeling progression will be used as the evaluation criterion.

Primary Objective:

The main goal is to demonstrate that mitral regurgitant volume assessed by 4DFlow-MRI is more strongly correlated with left ventricular (LV) remodeling progression after correction or persistence of MR than mitral regurgitant volume assessed by 2D MRI or TTE, after adjustment for residual MR.

The primary outcome criterion will be the analysis of the association between the absolute change in LV end-diastolic volume (LVEDV) between baseline (M0) and 6 months after (M6) and mitral regurgitant volume at M0, as calculated by the different methods or MR severity estimated using the integrative TTE approach, adjusted for residual MR.

Secondary Objectives:

1. Evaluate the association between LV remodeling and mitral regurgitant volume measured by the different methods in the subgroup of patients undergoing percutaneous intervention, where correction is incomplete and residual MR assessment is challenging.
2. Evaluate the association between LV remodeling and mitral regurgitant volume measured by the different methods in the subgroup of patients undergoing surgical intervention, where correction is expected to be excellent with no residual MR.
3. Analyze the determinants of LV remodeling progression using novel volumetric echocardiography methods, including specific ultrafast ultrasound sequences, allowing comparisons with data from the most innovative echocardiographic techniques.
4. Investigate all determinants of LV remodeling progression at six months beyond mitral regurgitant volume, including the significance of LV remodeling, longitudinal strains of the LV and left atrium (assessed by MRI and TTE), and myocardial fibrosis derived from myocardial T1 mapping before and after gadolinium injection at M0.

Secondary Outcomes Criteria:

1. Primary evaluation criterion assessed in the subgroup of patients who underwent percutaneous MR correction.
2. Primary evaluation criterion assessed in the subgroup of patients who underwent surgical MR correction, disregarding residual MR.
3. Primary evaluation criterion assessed using innovative echographic techniques, including specific ultrafast ultrasound sequences, and compared with the standard TTE, 2D MRI and 4D MRI.
4. Changes in LV remodeling between M0 and M6, based on various indices (LVEDV, fibrosis indices, strain at M0).

ELIGIBILITY:
Inclusion Criteria: Subjects

* from 18 to 85 years old
* having signed a consent form to participate in the study
* suffering from mild, moderate or severe mitral regurgitation based on an ultrasound graduation
* able to undergo echocardiography and IRM within 7 days after recruitment and then at 6 months

Exclusion Criteria: Subjects

* suffering from aortic regurgitation or stenosis or mitral stenosis associated with more than moderate MR, intracardiac shunting or hypertrophic cardiomyopathy
* suffering from secondary MR
* having a contraindication to gadolinium-based contrast agent
* having a pacemaker, defibrillator or any other contraindication to MRI
* suffering from renal disease with an eGFR CKD-EPI < 30 ml/min
* pregnant or breastfeeding
* under legal protection

Enrolled subjects:

* with an incomplete or suboptimal ultrasound or MRI examination
* who have not attended to the 6-month follow-up visit
* with an intercurrent medical event

will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Absolute change in left ventricle end-diastolic volume | Baseline, 6 months
  The primary outcome criterion will be the analysis of the association between the absolute change in LV end-diastolic volume (LVEDV) between baseline (M0) and 6 months after (M6) and mitral regurgitant volume at M0, as calculated by the different methods or MR severity estimated using the integrative TTE approach, adjusted for residual MR.
Mitral regurgitant volume | Baseline
  The primary outcome criterion will be the analysis of the association between the absolute change in LV end-diastolic volume (LVEDV) between baseline (M0) and 6 months after (M6) and mitral regurgitant volume at M0, as calculated by the different methods or MR severity estimated using the integrative TTE approach, adjusted for residual MR.

SECONDARY OUTCOMES:
Absolute change in left ventricle end-diastolic volume | Baseline, 6 months
  Same outcome as the primary outcome but in a subgroup of patients who have undergone percutaneous mitral regurgitation correction.
Mitral regurgitant volume | Baseline
  Same outcome as the primary outcome but in a subgroup of patients who have undergone percutaneous mitral regurgitation correction.
Absolute change in left ventricle end-diastolic volume | Baseline, 6 months
  Same outcome as the primary outcome but in a subgroup of patients who have undergone surgical mitral regurgitation correction.
Mitral regurgitant volume | Baseline
  Same outcome as the primary outcome but in a subgroup of patients who have undergone surgical mitral regurgitation correction.
Absolute change in left ventricle end-diastolic volume | Baseline, 6 months
  Same outcome as the primary outcome but mesured using ultrafast ultrasound imaging compared to the 3 other imaging techniques performed in the study.
Mitral regurgitant volume | Baseline
  Same outcome as the primary outcome but mesured using ultrafast ultrasound imaging compared to the 3 other imaging techniques performed in the study.
Change from baseline in left ventricle remodeling | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Soulat, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Groupe hospitalier Paris Saint-Joseph - hôpital Marie-Lannelongue, Le Plessis-Robinson
  - AP-HP - hôpital Saint-Antoine, Paris
  - AP-HP - hôpital européen Georges-Pompidou,, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).